CLINICAL TRIAL: NCT02800863
Title: TARGET: A Post-Approval Study to Evaluate Targeted SCS Spinal Cord Stimulation (SCS) Dorsal Root Ganglion (DRG) Stimulation for the Management of Moderate to Severe Chronic, Intractable, Pain of the Lower Limbs Due to CRPS Types I and II
Brief Title: TARGET Post-Approval Study
Acronym: TARGET PAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10113
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
Keywords: Complex Regional Pain Syndrome (CRPS); Chronic pain; SJM-CIP-10113
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dorsal Root Ganglion (DRG) Stimulation
  Interventions: Device: Dorsal Root Ganglion (DRG) Stimulation (Axium™ Neurostimulator System); Device: Dorsal Root Ganglion (DRG) Stimulation (Proclaim™ Neurostimulator System)

INTERVENTIONS:
Device: Dorsal Root Ganglion (DRG) Stimulation (Axium™ Neurostimulator System) — Electrical stimulation of the DRG using the Axium™ Neurostimulator System
Device: Dorsal Root Ganglion (DRG) Stimulation (Proclaim™ Neurostimulator System) — Electrical Stimulation of the DRG using the Proclaim™ Neurostimulator System.

SUMMARY:
The purpose of this prospective, multicenter, single arm post-approval study is to demonstrate continued safety of the Axium and Proclaim Neurostimulator System for dorsal root ganglion (DRG) stimulation. The primary endpoint is the 12-month serious adverse event rate for permanent implants.

DETAILED DESCRIPTION:
A maximum of 426 adult subjects with moderate to severe chronic, intractable, pain of the lower limbs due to CRPS types I and II will undergo a trial of the Axium or Proclaim Neurostimulator System across up to 45 study sites in the United States. Only subjects who report a 50% or greater reduction in overall pain intensity through direct patient-reported percentage of pain relief will receive the permanent implant. Subjects will then return to the office for follow-up at 1, 3, 6 and 12 months post-permanent implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between ≥ 22 and ≤ 75 years of age.
* Subject has moderate to severe chronic intractable pain of the lower limbs resulting from Complex Regional Pain Syndrome (CRPS) types I or II.
* Subject has a baseline Visual Analogue Scale (VAS) of ≥ 60 mm for overall pain at the time of the baseline assessment.
* Subject is willing and able to comply with the study requirements.
* Subject is able to provide written informed consent.

Exclusion Criteria:

* Subject has an active implantable medical device including but not limited to cardiac pacemakers and cardiac defibrillators.
* Subject is currently involved in medically related litigation, including workers compensation.
* Subject has a life expectancy of less than one year.
* Subject is pregnant or of child bearing potential and not using adequate contraception as determined by the investigator.
* Subject has, or plans to have, a spinal cord stimulation system or infusion pump system implanted.
* Subject has, or plans to have, a peripheral nerve stimulation system (PNS) or peripheral nerve field stimulation system (PNfS) implanted.
* Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the implant procedure and/or recovery from the implant procedure or could complicate the required procedures and evaluations of the study in the judgment of the investigator.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects aged 22 to 75 with moderate to severe chronic, intractable, pain of the lower limbs due to CRPS types I and II with a baseline VAS score of 6 or greater.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Jannu, PhD, CCRP, Study Director — Abbott Neuromodulation
Locations (44):
- United States (44):
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Spanish Hills Interventional Pain Specialists, Camarillo, California
  - California Orthopedics & Spine, Larkspur, California
  - Loma Linda University Hospital, Loma Linda, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - University of California - San Francisco, San Francisco, California
  - Orthopedic Pain Specialists, Santa Monica, California
  - Summit Pain Alliance Inc., Santa Rosa, California
  - Pacific Research Institute, Santa Rosa, California
  - Front Range Pain Medicine, Fort Collins, Colorado
  - Coastal Orthopedics & Sports Medicine Southwest FL, Bradenton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida - Department of Anesthesia, Gainesville, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - Better Health Clinical Research, Newnan, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Goodman Campbell Brain & Spine, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Nura, Edina, Minnesota
  - Twin Cities Pain Clinic, Edina, Minnesota
  - Advanced Pain Care, Henderson, Nevada
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Ainsworth Institute of Pain Management, New York, New York
  - The Spine & Pain Institute of New York, Staten Island, New York
  - Premier Pain Solutions, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Adena Bone and Joint Center, Chillicothe, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Pacific Sports and Spine, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Spinal Diagnostics, Tualatin, Oregon
  - Center for Intervetional Pain and Spine, Exton, Pennsylvania
  - Main Line Spine, King of Prussia, Pennsylvania
  - Thomas Jefferson Department of Neurosurgery, Philadelphia, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Carolinas Center for Advanced Management of Pain, Greenville, South Carolina
  - Vertex Spine and Pain, Franklin, Tennessee
  - Central Texas Pain Institute, Killeen, Texas
  - Advanced Pain Solutions, Mesquite, Texas
  - Shannon Clinic, San Angelo, Texas
  - The Spine and Nerve Center of St. Francis, Charleston, West Virginia
  - Advanced Pain Management, Greenfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 426 subjects at 44 investigational sites. The first subject was enrolled in August 2016 and the last subject in December 2019. Completion of enrollment and follow-up in the study occurred in September 2021.
Period: Overall Study
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Started | 426
Completed | 198
Not Completed | 228
Not completed — Adverse Event | 14
Not completed — Another Device Implanted | 1
Not completed — Device Explanted | 1
Not completed — Device Has Been Turned Off Since Jan 2019 | 1
Not completed — Health Issues | 1
Not completed — Insurance Denial | 8
Not completed — No Perm Implant, Active Pain Pump Implanted | 1
Not completed — Patient Did not Obtain at Least 50% Pain Relief | 1
Not completed — Screen Failure | 1
Not completed — Sponsor Request | 6
Not completed — Death | 3
Not completed — Subject Implant at Another Facility | 1
Not completed — Lost to Follow-up | 26
Not completed — Subject Participation Terminated by Investigator | 17
Not completed — Subject and/or Family Request | 64
Not completed — Trial Failure | 81
Not completed — Used Different Battery not Approved for Study at Time of Perm | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Number analyzed (Participants) | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259
  Male | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 375
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 361
  More than one race | 17
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 426
Complex Regional Pain Syndrome (CRPS) [Count of Participants; unit: Participants] — Subject has moderate to severe chronic intractable pain of the lower limbs resulting from Complex Regional Pain Syndrome (CRPS) types I or II.
  Type I occurs when there is no confirmed nerve injury. Type II is when there is known associated nerve injury. The enrolling physicians diagnosed the CRPS type.
  Participants
    CRPS I | 301
    CRPS II | 125

OUTCOME MEASURES:

1. Primary Outcome: Rate of Serious Adverse Events (SAEs)
Description: The serious adverse event rate for subjects receiving the permanent DRG implantable pulse generator (IPG) was analyzed using Kaplan-Meier method on subjects who received the permanent Axium or Proclaim DRG IPG (N = 296). While 426 patients were enrolled, only 296 received the permanent implant. The primary population is 296.
Time Frame: throughout 12 month study
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Error); unit: percentage of events
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Number analyzed (Participants) | 296
percentage of events | 8.7 (1.7)

2. Secondary Outcome: Percent Change From Baseline to 12 Months Post-permanent Implant for Overall Pain Intensity Measured Using the Visual Analog Scale (VAS)
Description: The VAS is a common, self-administered measure in which subjects rate their pain intensity by marking a vertical line through a 100 mm horizontal line anchored by word descriptors on each end (no pain to worst imaginable pain). The distance between the beginning of the horizontal line and the vertical line is measured to produce a score between 0 and 100 mm (or 0 to 10 cm). A higher score indicates higher pain intensity and a 30% reduction in VAS score from baseline to follow-up is considered clinically relevant.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Number analyzed (Participants) | 213
percent | 44.48 (34.15)

3. Secondary Outcome: Change From Baseline to 12 Months Post-permanent Implant for Physical Function Measured Using the Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) Physical Function Scale
Description: The PROMIS-29 Profile is an instrument made up of seven individual short forms (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference) that are scored individually. The instrument also includes a single pain intensity item which is reported as its raw score (e.g., 0 to 10). Each item has five response options ranging in value from 1 to 5, except for the Pain Intensity item which has eleven response options ranging in value from 0 to 10. A raw score is created from each short form that makes up the Profile. Raw scores are calculated by summing the values of the response to each question within each domain.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Number analyzed (Participants) | 212
percent | 5.13 (6.28)

4. Secondary Outcome: Change From Baseline to 12 Months Post-permanent Implant for Quality of Life Measured Using the PROMIS Global Health Scale
Description: The PROMIS Global Health short form is a validated, 10-item instrument designed to assess multiple health domains. The questionnaire yields a total score and sub-scale scores for Global Physical and Mental Health. Each question has potential five response options ranging in value from one to five to give a total score ranging from 10 to 50. All questions must be answered to arrive at a total score as one or more missing responses will render scores unusable. Scores are converted into t-scores where the average for the general US population is 50 and the SD is 10. Higher scores indicate better global health.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
Number analyzed (Participants) | 426
percent
  Physical Health: number analyzed (Participants) | 219
  Physical Health | 6.22 (7.25)
  Mental Health: number analyzed (Participants) | 218
  Mental Health | 4.42 (8.19)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Dorsal Root Ganglion (DRG) Stimulation
All-Cause Mortality (participants affected / at risk) | 3/426
Serious Adverse Events (participants affected / at risk) | 26/426
Other Adverse Events (participants affected / at risk) | 5/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dorsal Root Ganglion (DRG) Stimulation (N=426)
Cellulitis (Infections and infestations) | 1
Acute Community Acquired Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Altered Mental Status (Psychiatric disorders) | 1
Ankle Surgery (Surgical and medical procedures) | 1
Bone Fracture (General disorders) | 1
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular Accident (Vascular disorders) | 1
Chest Pain (General disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 1
Covid Associated Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Crohns Disease Flare Up (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Dizziness and Chest Pain (General disorders) | 1
Embolism (General disorders) | 2
Epistaxis (General disorders) | 1
Escalating Pain (General disorders) | 1
Fall (General disorders) | 1
Gastrointestinal or Genitourinary Compromise (Gastrointestinal disorders) | 2
Infection (Infections and infestations) | 1
Infection in Foot (Infections and infestations) | 1
Knee Infection (Infections and infestations) | 1
Myocardial Infarction (Cardiac disorders) | 1
Numbness (General disorders) | 1
Patient Had Sub-Acute CVA 7 Days After Trial (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5
Right Ankle Fracture (General disorders) | 1
Sepsis (Infections and infestations) | 1
St Elevation Myocardial Infarction (Cardiac disorders) | 1
Toe Amputation (General disorders) | 1
Unrelated Trauma (General disorders) | 1
Vertebral Compression Fracture (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dorsal Root Ganglion (DRG) Stimulation (N=426)
Clumsiness (General disorders) | 2
Dizziness (General disorders) | 1
Pain at the Implant Site (Injury, poisoning and procedural complications) | 1
Tibial Nerve Surgery (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor Review. Principal investigator and Institution shall provide a copy of any abstract, presentation, journal, manuscript (written by Principal Investigator or Study Staff) and all related materials relating to the Study to Sponsor at least sixty (60) days prior to the proposed submission date.

DOCUMENTS (2):
  • Study Protocol (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02800863/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02800863/SAP_001.pdf